CLINICAL TRIAL: NCT07105163
Title: Observational, Cross-sectional, Multicenter Study to Evaluate Adherence to Different Treatment Regimens With Oral Bisphosphonates and Calcium and Vitamin D Supplements in Postmenopausal Osteoporosis.
Brief Title: Evaluation of Adherence With Bisphosphonates and Calcium and Vitamin D Supplements in Women With Postmenopausal Osteoporosis
Acronym: OSTEOAD
Status: Recruiting | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: OSTEOAD
Record Dates: First submitted 2025-06-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Post Menopausal Osteoporosis
Keywords: Procare; Post menopausal osteoporosis; Bisphosphonate; calcium; vitamin D; supplement
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the adherence of patients to combined treatment with bisphosphonates and calcium and vitamin D supplements, which is one of the usual treatments for postmenopausal osteoporosis. The study will consist of a single visit that will coincide with one of the patient's usual follow-up visits according to standard clinical practice. During this visit, information will be collected from the patient's medical history and an interview will be conducted using 3 questionnaires to assess how and how often the patient takes the treatment, possible forgetfulness, and whether or not the patient is satisfied with their current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. - Women diagnosed with postmenopausal OP.
2. - Women who had been prescribed oral treatment with a BP administered monthly or weekly together with a Ca/D supplement (sachets or chewable tablets) administered daily, at least 6 months prior to inclusion in the study.
3. - Women who had given their written informed consent before participating in the study.

Exclusion Criteria:

None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with postmenopausal osteoporosis who have been prescribed treatment with an oral bisphosphonate combined with Ca/D supplements.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intergroup adherence | Day 1
  To evaluate intergroup adherence to the most common oral regimens used in the treatment of postmenopausal OP that combine BP and Ca/D supplements, using a 8-items Morisky Medication Adherence Scale

SECONDARY OUTCOMES:
Persistence intergroup | Day 1
  To evaluate, intergroup, the persistence to the most common oral regimens used in the treatment of postmenopausal OP that combine BP and Ca/D supplements. It will be evaluated over time from the start of the combination of both until the first end date of administration of either one, and by the percentage of patients who continue with the combined treatment since its prescription
Adherence intragroup | Day 1
  To evaluate, intragroup, the adherence to the prescribed usual oral regimens, using a 8-items Morisky Medication Adherence Scale
Persistence intragroup | Day 1
  To evaluate, intragroup, the persistence to the prescribed usual oral regimens.
Factors of non-adherence | Day 1
  To evaluate possible determining factors of non-adherence to the prescribed usual oral regimens and their comparison between the different regimens.
Factors of non-persistence | Day 1
  To evaluate possible determining factors of non-persistence to the prescribed usual oral regimens and their comparison between different regimens.
Treatment satisfaction | Day 1
  To evaluate the patient's satisfaction with the combined treatment received using a Likert scale.

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Clinica Gaias Santiago, Santiago de Compostela, A coruña
  - CP Dr Caracuel, Córdoba, Andalusia
  - Hospital Reina Sofia, Córdoba, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - CP Dr Agramonte, Palma de Mallorca, Balearic Islands
  - CP Dr Balta, Palma de Mallorca, Balearic Islands
  - CHU Insular - H Materno-Infantil, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Zamora, Zamora, Castille and León
  - Clinica Sagrada Familia, Barcelona, Catalonia
  - CP Dra Sanchez, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital del Tajo, Aranjuez, Madrid
  - CP Dr Solano, Madrid, Madrid
  - CP Dr Zafra, Madrid, Madrid
  - CP Dra Gerechter, Madrid, Madrid
  - Hospital Infanta Leonor, Madrid, Madrid
  - Hospital Virgen del Mar, Madrid, Madrid
  - CP Dr Larrauri, Vigo, Pontevedra
  - CP Dra Medrano, Alicante, Valencia
  - CP Dra Tejon, Alicante, Valencia

IPD SHARING:
Plan to Share IPD: No